CLINICAL TRIAL: NCT02707328
Title: Phase I Study To Establish Maximum Tolerated Dose (MTD) of Cyberknife in Patients With Un-Resectable Pancreas Cancer (TL002)
Brief Title: Study To Establish Maximum Tolerated Dose (MTD) of Cyberknife in Patients With Un-Resectable Pancreas Cancer (TL002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed after being on administrative hold
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-176
Record Dates: First submitted 2015-10-02; First posted 2016-03-14 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Adenocarcinoma of the Pancreas; Pancreas Adenocarcinoma; Pancreatic Adenocarcinoma
Keywords: Gemcitabine; Gemzar; CyberKnife; Cyber knife; CK; abraxane; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Chemotherapy:
  Gemcitabine 1000 mg/m2 and Abraxane 125 mg/m2 weekly x3 of 28 day cycle
  Radiation:
  20-55 GY over 5 fractions
  Dosing schedule: 3 cycles of chemotherapy, followed by CyberKnife, followed by 3 additional cycles of chemotherapy.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Radiation: CyberKnife

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: gemzar
Drug: nab-paclitaxel
  Other Names: abraxane
Radiation: CyberKnife
  Other Names: cyber knife, CK, Stereotactic radiosurgery

SUMMARY:
This study is looking at determining the maximum safe dose of CyberKnife when given with chemotherapy for unresectable adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
The purpose of this study is to determine the MTD for radiosurgery in the treatment of unresectable pancreas cancer, this MTD can then be used in future phase II or III studies. In terms of starting dose for the phase I study, based on the low toxicity seen in the Moffitt study we feel that 30 Gy in five fractions will be a successful starting dose.

Most of the data in unresectable is derived from patients in the metastatic setting in terms of chemotherapy agents. There have been two major studies that looked at various chemotherapy regimens versus the previous standard of care Gemzar. One study found improved survival with FOLFIRINOX and a second found that the combination of nab-paclitaxel and gemzar were superior to gemzar alone. Thus, the current standard of care for metastatic pancreas cancer (in which a local therapy like radiation has more limited role) is either FOLFIRINOX or gemzar and nab-paclitaxel. While there is some discussion of a randomized study comparing FOLFIRINOX and gemzar combined with nab-paclitaxel such a study has not started as of this time and it is unclear how much interest there would be in accruing to this study. Therefore the exact best chemotherapy regimen for metastatic disease is unclear but is either FOLFIRIONX or gemzar-nab-paclitaxel. The chemotherapy regimens for unresectable cancer are extrapolated from the metastatic setting, per NCCN guidelines any chemotherapy regimen approved for metastatic disease is reasonable to use in unresectable pancreas cancer. Thus for purpose of this study we have chosen one of the two chemotherapy regimens that have shown the best results in the metastatic setting, since there is no way to determine the exact best regimen we have chosen gemzar and nab-paclitaxel since it is felt that this is a less toxic regimen as compared to FOLFIRINOX.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas
* Unresectable disease based on the following imaging criteria (table 1)

  * extrapancreatic extension
  * tumor involvement of the SMA or celiac axis
  * evidence of occlusion of the SMV-portal vein confluence
* KPS > 50 (ECOG 0-2)
* Age >18 years
* Women of childbearing age and male participants must practice adequate contraception (hormonal or barrier method of birth control; abstinence) prior to and throughout study treatment.
* Life expectancy > 3 months
* Ability to understand and the willingness to sign a written informed consent.
* Note that patients with metastatic disease are eligible if it is felt that the patients will benefit from local control of the primary disease.
* Disease that is measureable or evaluable for response endpoint per RECIST

Exclusion Criteria:

* Prior radiotherapy to the upper abdomen
* Resectable or borderline resectable pancreas cancer. Note that these patients are eligible for a separate study looking at radiosurgery for borderline resectable pancreas cancer
* Severe comorbidity rendering a candidate ineligible for chemotherapy or radiation, Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients of childbearing age who are unwilling or unable to practice contraception
* Inability to undergo MRI or CT with contrast for treatment planning
* Patients may not be receiving any other investigational nor commercial agents with therapeutic intent to treat pancreatic cancer while on this trial. Note that patients can have had previous investigational therapy but cannot have this concurrently with this protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose | 4-7 months
  This study is to evaluate the MTD for Cyberknife when given in conjunction with Gemcitabine and Abraxane.

SECONDARY OUTCOMES:
overall survival | 6 months, 1 year, 5 years
Tumor response per RECIST 1.1 | 4 months, 6 months, 1 year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 months, 6 months, 1 year
quality of life | 2 months, 4 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center at Cooper, Camden, New Jersey, United States